CLINICAL TRIAL: NCT06549023
Title: Single Session vs Multiple-Session Panretinal Photocoagulation With Navigated Laser in Proliferative Diabetic Retinopathy - The SMART-PRP Study
Brief Title: Single Session vs Multiple-Session Panretinal Photocoagulation for Treatment of Proliferative Diabetic Retinopathy
Acronym: SMART-PRP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vastra Gotaland Region (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SMART-PRP
Record Dates: First submitted 2024-08-08; First posted 2024-08-12 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-10

CONDITIONS: Proliferative Diabetic Retinopathy; Diabetic Retinopathy; Diabetic Retinopathy Visually Threatening; Diabetic Macular Edema; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2
Keywords: Panretinal photocoagulation (PRP); Single-session PRP; Multiple-session PRP; Navigated laser; Navilas; Central subfield retinal thickness (CRT); Macular volume; Optical coherence tomography (OCT); Swept-source optical coherence tomography (SS-OCT); Wide-field fundus imaging; OCT-angiography; Retinal oximetry; Electroretinogram (ERG)
MeSH Terms: conditions — Diabetic Retinopathy; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: Participants will be randomly allocated to either the single-session (SS-PRP) or multiple-sessions (MS-PRP) panretinal photocoagulation groups using a computer-generated sequence. Block randomization will be utilized to ensure balanced group sizes and comparable participant characteristics.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Single-session panretinal PRP (SS-PRP) (Active Comparator): Administration of all panretinal photocoagulation (PRP) treatment in one comprehensive session, typically delivered in a single clinical visit.
  Interventions: Procedure: Single-session panretinal PRP (SS-PRP)
- Multiple-session panretinal PRP (MS-PRP) (Active Comparator): Administration of panretinal photocoagulation (PRP) treatment over two separate visits with at least one week apart.
  Interventions: Procedure: Multiple-session panretinal PRP (MS-PRP)

INTERVENTIONS:
Procedure: Single-session panretinal PRP (SS-PRP) — Administration of panretinal photocoagulation (PRP) treatment with navigated laser using Navilas in one comprehensive session, typically delivered in a single clinical visit.
  Arms: Single-session panretinal PRP (SS-PRP)
Procedure: Multiple-session panretinal PRP (MS-PRP) — Administration of panretinal photocoagulation (PRP) treatment with navigated laser using Navilas over two separate visits with at least one week apart.
  Arms: Multiple-session panretinal PRP (MS-PRP)

SUMMARY:
Proliferative diabetic retinopathy (PDR) is the leading cause for blindness in working-age adults. The current gold standard treatment for PDR is panretinal photocoagulation (PRP). In current clinical practice, both single-session and multiple-session PRP approaches are widely accepted and utilized. The purpose of this study is to compare the safety and effectiveness of single-session and multiple-session PRP.

DETAILED DESCRIPTION:
Proliferative diabetic retinopathy (PDR) is a well-known complication for both type 1 and type 2 diabetes mellitus (DM) and it is the leading cause for blindness in working-age adults. The current gold standard treatment for PDR, established more than four decades ago by the Diabetic Retinopathy Study (DRS), is panretinal photocoagulation (PRP). The treatment goal is to halt the progression of PDR by destroying parts of the peripheral retina in a pattern fashion and hence preserving the visually important central macular region. The tissue destruction reduces the area of ischemia and reduces the production of vascular endothelial growth factor (VEGF), which drives the formation of neovascular proliferations. In the management of PDR, panretinal photocoagulation (PRP) stands as a cornerstone treatment. In current clinical practice, both single-session and multiple-session PRP approaches are widely accepted and utilized. The choice between these approaches often depends on the practitioner's preference, patient characteristics, and specific clinical circumstances.

Although both single-session and multiple-session PRP are employed in practice, there's an ongoing debate regarding their comparative safety and effectiveness. Older studies suggest a heightened risk of diabetic macular edema (DME) with single-session PRP, while newer research, particularly those involving milder laser techniques, indicates that the risk might be similar regardless of the number of sessions. This inconsistency in findings underscores the need for further research and the investigators aim to shed light over this with this prospective, controlled and randomized interventional study.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years.
* Patients with type 1 or type 2 Diabetes Mellitus with newly diagnosed Proliferative Diabetic Retinopathy, PDR.
* Visual acuity ≥ 0.1 Snellen.
* CRT of less than 300 micrometer measured by OCT without cysts in the neuroretina.
* Clear media and adequately dilated pupil for PRP.

Exclusion Criteria:

* Intraocular surgery within the last 4 months or planned within the next 3 months.
* Previous or current center-involved diabetic macular edema (Ci-DME).
* Previous PRP, intravitreal treatment (IVT), or macular laser treatment in study eye.
* Treatment with medications known to risk macular edema.
* Media opacity preventing adequate PRP.
* General medical condition making office laser treatment very difficult or impossible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Central subfield retinal thickness (CRT) | Baseline and 1, 3 and 6 months after treatment
  Mean change from baseline in CRT
Vessel Perfusion Density (VPD) | Baseline and 1, 3 and 6 months after treatment
  Mean change from baseline in VPD
Vessel Length Density (VLD) | Baseline and 1, 3 and 6 months after treatment
  Mean change from baseline in VLD
Foveal Avascular Zone (FAZ) | Baseline and 1, 3 and 6 months after treatment
  Mean change from baseline in FAZ
Lesion size | Baseline and 1, 3 and 6 months after treatment
  Mean change from baseline in lesion size
Macular volume | Baseline and 1, 3 and 6 months after treatment
  Mean change from baseline in macular volume
Venular saturation | Baseline and 1, 3 and 6 months after treatment
  Mean change from baseline in venular saturation
Arteriolar saturation | Baseline and 1, 3 and 6 months after treatment
  Mean change from baseline in arteriolar saturation
Retinal diameter | Baseline and 1, 3 and 6 months after treatment
  Mean change from baseline in retinal diameter
Venular diameter | Baseline and 1, 3 and 6 months after treatment
  Mean change from baseline in venular diameter
Retinal function | Baseline and 1, 3 and 6 months after treatment
  Mean change from baseline in retinal function using full-field electroretinogram (ERG)
Diabetic macular edema (DME) | Baseline and 1, 3 and 6 months after treatment
  Incidence of diabetic macular edema (DME)
Subjective experience of pain after treatment | Baseline and 1, 3 and 6 months after treatment
  Study patients' subjective experience of pain after treatment using visual analog scale (VAS)
Subjective overall experience of the treatment | Baseline and 1, 3 and 6 months after treatment
  Study patients' subjective overall experience of the treatment using verbal scale (VS)
Cost-effectiveness | Baseline and 1, 3 and 6 months after treatment
  We intend to conduct a thorough cost-effectiveness analysis, comparing the single-session approach with the traditional multiple-session treatments.
  This analysis will factor in direct medical costs, including the expenses related to the laser equipment, healthcare professionals' time, and the required clinical facilities. We will also consider indirect costs such as patient travel expenses and time taken off work.

CONTACTS AND LOCATIONS:
Overall Officials: Marita Andersson Grönlund, M.D. Prof, Principal Investigator — Göteborg University
Locations (1):
- Ögonmottagning Mölndal/SU, Mölndal, Sweden